CLINICAL TRIAL: NCT07231991
Title: A PHASE 1, NON-RANDOMIZED, OPEN-LABEL, SINGLE-DOSE, PARALLEL GROUP STUDY TO COMPARE THE PHARMACOKINETICS OF VEPDEGESTRANT (PF-07850327) IN ADULT PARTICIPANTS WITH MODERATE AND SEVERE HEPATIC IMPAIRMENT RELATIVE TO HEALTHY PARTICIPANTS WITH NORMAL HEPATIC FUNCTION
Brief Title: A Study to Learn How the Body Processes the Study Medicine Called Vepdegestrant in People With Loss of Liver Function
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arvinas Estrogen Receptor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C4891004
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): participants with normal hepatic function
  Interventions: Drug: vepdegestrant
- Group 2 (Experimental): participants with moderate hepatic impairment
  Interventions: Drug: vepdegestrant
- Group 3 (Experimental): participants with severe hepatic impairment
  Interventions: Drug: vepdegestrant

INTERVENTIONS:
Drug: vepdegestrant — Vepdegestrant administered as a single oral 200 mg dose
  Other Names: ARV-471, PF-07850327

SUMMARY:
The purpose of the study is to look at how the body processes a study medicine called vepdegestrant in participants with loss of liver function relative to people with normal liver function.

This study is seeking participants who are:

* females who cannot have children or males
* between 18 and 70 years of age
* weigh more than 50 Kilograms (110 pounds)
* either healthy with normal liver function or have loss of liver function

All participants in this study will take one dose of vepdegestrant by mouth. This study looks at how the medicine is changed and removed from the body after being taken by the participants. The amount of vepdegestrant in participants with loss of liver function will be compared to the amount of vepdegestrant in participants with normal liver function.

All participants will stay at the study clinic for about 11 days and 10 nights.

ELIGIBILITY:
Inclusion criteria including but not limited to:

* Female participants of non-childbearing potential, or male participants between the age of 18 years (or the minimum age of consent in accordance with local regulations) and 70 years, inclusive, at screening.
* Body mass index of 17.5-38 kg/m2, inclusive, and a total body weight >50 kg (110 lb).

Normal hepatic function group only:

-Overtly healthy as determined by medical evaluations including medical history, physical examination, laboratory tests, vital signs and standard 12-lead ECGs.

Hepatic impairment groups only:

* Satisfy the criteria for Class B (Group 2: moderate hepatic impairment) or C (Group 3: severe hepatic impairment) of the modified Child-Pugh Classification.
* Stable hepatic impairment, defined as no clinically significant change in disease status within the last 28 days prior to the screening visit, as documented by the participant's recent medical history.

Exclusion criteria including but not limited to:

* Any condition possibly affecting drug absorption.
* Use of prohibited prior or concomitant medications.

Normal hepatic function group only:

-Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

Hepatic impairment groups only:

-A diagnosis of hepatic dysfunction secondary to any acute ongoing hepatocellular process that is documented by medical history, PE, liver biopsy, hepatic ultrasound, CT scan, or MRI.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11-04 (Estimated); Primary Completion 2026-11-29 (Estimated); Study Completion 2026-12-23 (Estimated)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) for vepdegestrant | Pre-dose, and 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 96, 120, 144, 168, 192, and 216 hours post dose
Area under the curve from time zero to extrapolated infinite time [AUC (0 - ∞)] for vepdegestrant | Pre-dose, and 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 96, 120, 144, 168, 192, and 216 hours post dose
  AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).

SECONDARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events | Time from baseline through and including follow-up contact occurring 28 to 35 calendar days after the last administration of the study intervention.
Number of Participants With Clinically Significant Clinical Laboratory Abnormalities | Time from baseline through and including follow-up contact occurring 28 to 35 calendar days after the last administration of the study intervention.
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Time from baseline through and including follow-up contact occurring 28 to 35 calendar days after the last administration of the study intervention.
Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities | Time from baseline through and including follow-up contact occurring 28 to 35 calendar days after the last administration of the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4891004